CLINICAL TRIAL: NCT06398223
Title: Ocular Perfusion in Patients With Unilateral Carotid Artery Stenosis
Status: Recruiting | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Assoc. Prof. Priv. Doz. Dr. med. univ., Medical University of Vienna
Other Study IDs: OPHT-101023
Record Dates: First submitted 2024-04-22; First posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Carotid Artery Stenosis
MeSH Terms: conditions — Carotid Stenosis | interventions — Endarterectomy, Carotid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Carotid endarterectomy (CEA) (Group 1): Subjects with unilateral carotid artery stenosis and planned CEA
  Interventions: Procedure: Carotid endarterectomy (CEA)
- Carotid artery stenting (Group 2): Subjects with unilateral carotid artery stenosis and planned carotid artery stenting
  Interventions: Procedure: Carotid artery stenting
- Healthy Control Group (Group 3): Healthy age- and sex-matched control subjects

INTERVENTIONS:
Procedure: Carotid endarterectomy (CEA) — Carotid endarterectomy (CEA): Surgical procedure to remove the plaque buildup in the carotid artery.
  Groups: Carotid endarterectomy (CEA) (Group 1)
Procedure: Carotid artery stenting — Carotid artery stenting: Treatment of the stenosis with a stent. The plaque in the artery wall is not removed but the narrowing is dilated.
  Groups: Carotid artery stenting (Group 2)

SUMMARY:
The aim of the presented study is to evaluate ocular blood flow, respectively optic nerve head blood flow in patients with carotid artery stenosis before and after carotid endarterectomy or carotid artery stenting. Additionally, the investigators aim to compare optic nerve head blood flow in patients with CAS and healthy age- and sex-matched control subjects. Furthermore, the investigators intend to evaluate brain tissue oxygenation in patients with carotid artery stenosis before, during and after CEA and carotid artery stenting. Finally, the investigators will assess potential correlations between LSFG and NIRS results in patients with unilateral carotid artery stenosis.

DETAILED DESCRIPTION:
Carotid artery stenosis is a condition that can lead to severe consequences such as ocular ischemia or stroke. As the ophthalmic artery branches off the carotid artery, ocular ischemic complications include amaurosis fugax, ocular ischemic syndrome or central retinal artery occlusion. Hence, early diagnosis of carotid artery stenosis and ocular perfusion impairment is of considerable importance to prevent ocular and systemic ischemic complications.

As the retina offers a unique window for examining the microcirculation in a non-invasive manner, several imaging techniques have already been used in recent years to assess ocular alterations associated with carotid artery stenosis. However, these examination techniques have their limitations and are therefore not suitable methods for determining ocular perfusion. On the contrary, Laser Speckle Flowgraphy (LSFG) is a non-invasive, in-vivo imaging method which quantitatively estimates blood flow in the optic nerve head, the choroid, the retina and the iris. LSFG offers a promising alternative from conventional methods, as it eliminates the need for contrast agents, has a low procedural complexity and obtains precise and reproducible measurements.

As the eye and brain share a close vascular relationship, both receiving blood supply from branches of the internal carotid artery, there is potential to establish a correlation between cerebral and ocular hemodynamics. Near-infrared spectroscopy (NIRS) is a simple and non-invasive method which enables continuous assessment of cerebral oxygenation. However, data on the course of oxygenation of the brain tissue using NIRS before, during and after carotid interventions are scarce. Additionally, there is a lack of comparative NIRS data between carotid endarterectomy (CEA) and carotid artery stenting. Furthermore, correlation studies between oxygenation of the brain tissue and ocular perfusion are largely missing.

Hence, the aim of this study is to evaluate optic nerve head blood flow in patients with carotid artery stenosis before and after CEA or carotid artery stenting. Additionally, the investigators will compare optic nerve head blood flow in patients with carotid artery stenosis to healthy sex- and age-matched control subjects. Furthermore, the investigators intend to evaluate brain tissue oxygenation in patients with carotid artery stenosis before, during and after CEA and carotid artery stenting. Finally, the investigators will assess potential correlations between LSFG and NIRS results in patients with unilateral carotid artery stenosis.

ELIGIBILITY:
Inclusion Criteria for patients with unilateral carotid artery stenosis:

* Men and Women aged ≥ 18 years
* Signed informed consent
* Normal ophthalmic findings, unless the investigator considers an abnormality to be clinically irrelevant
* Diagnosis of unilateral carotid artery stenosis and scheduled carotid endarterectomy or carotid artery stenting

Inclusion criteria for healthy age- and sex-matched control subjects:

* Men and Women aged ≥ 18 years
* Signed informed consent
* Normal ophthalmic findings, unless the investigator considers an abnormality to be clinically irrelevant
* Normal findings in the medical history, unless the investigator considers an abnormality to be clinically irrelevant
* Non-Smokers

Exclusion criteria for patients with carotid artery stenosis and healthy age- and sex-matched control subjects:

* Blood donation in the three weeks preceding the study
* Symptoms of a clinically relevant illness in the three weeks preceding the study
* Ocular inflammation or infection within the last 3 months
* History of family history of epilepsy
* Diabetes mellitus type 1 or type 2
* Pregnant or breast-feeding women
* Women of childbearing potential (neither menopausal, nor hysterectomized, nor sterilized) not using effective contraception

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A total of 45 patients will be included in the study:
  * 15 subjects with unilateral carotid artery stenosis and planned CEA
  * 15 subjects with unilateral carotid artery stenosis and planned carotid artery stenting
  * 15 healthy age- and sex-matched control subjects
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2024-04-09 (Actual); Primary Completion 2026-05-02 (Estimated); Study Completion 2026-05-02 (Estimated)

PRIMARY OUTCOMES:
Optic nerve head blood flow | Before and 4-6 weeks after CEA or carotid artery stenting
  Change in optic nerve head blood flow (LSFG) in patients with unilateral carotid artery stenosis before and after carotid endarterectomy or carotid artery stenting

SECONDARY OUTCOMES:
Retinal oxygen saturation and retinal vessel diameter | Before and 4-6 weeks after CEA or carotid artery stenting
  Change in retinal oxygen saturation and retinal vessel diameter (retinal oximetry)

OTHER OUTCOMES:
Neurovascular coupling | Before and 4-6 weeks after CEA or carotid artery stenting
  Change in neurovascular coupling (retinal stimulation with flickering-light)
Retinal nerve fiber layer thickness | Before and 4-6 weeks after CEA or carotid artery stenting
  Change in retinal nerve fiber layer thickness (OCT)
Retinal thickness | Before and 4-6 weeks after CEA or carotid artery stenting
  Change in retinal thickness (OCT)
Retinal vessel density | Before and 4-6 weeks after CEA or carotid artery stenting
  Change in retinal vessel density (OCT-A)
Choroidal vascularity index | Before and 4-6 weeks after CEA or carotid artery stenting
  Change in choroidal vascularity index (EDI-OCT)
Optic nerve head blood flow | Before and 4-6 weeks after CEA or carotid artery stenting
  Change in optic nerve head blood flow (LDF)
OPP and arterial BP | Before and 4-6 weeks after CEA or carotid artery stenting
  Change in ocular perfusion pressure and arterial blood pressure
Brain tissue oxygenation | Before and 4-6 weeks after CEA or carotid artery stenting
  Change in brain tissue oxygenation (NIRS) before, during and after CEA or carotid artery stenting
NIRS and LSFG | Before and 4-6 weeks after CEA or carotid artery stenting
  Correlation between optic nerve head blood flow and brain tissue oxygenation before and after CEA or carotid artery stenting (LSFG and NIRS)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clincal Pharmacology, Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Background] Ismail A, Ravipati S, Gonzalez-Hernandez D, Mahmood H, Imran A, Munoz EJ, Naeem S, Abdin ZU, Siddiqui HF. Carotid Artery Stenosis: A Look Into the Diagnostic and Management Strategies, and Related Complications. Cureus. 2023 May 9;15(5):e38794. doi: 10.7759/cureus.38794. eCollection 2023 May. PMID 37303351
- [Background] Lahme L, Marchiori E, Panuccio G, Nelis P, Schubert F, Mihailovic N, Torsello G, Eter N, Alnawaiseh M. Changes in retinal flow density measured by optical coherence tomography angiography in patients with carotid artery stenosis after carotid endarterectomy. Sci Rep. 2018 Nov 21;8(1):17161. doi: 10.1038/s41598-018-35556-4. PMID 30464189
- [Background] Pierro L, Arrigo A, De Crescenzo M, Aragona E, Chiesa R, Castellano R, Catenaccio B, Bandello F. Quantitative Optical Coherence Tomography Angiography Detects Retinal Perfusion Changes in Carotid Artery Stenosis. Front Neurosci. 2021 Apr 22;15:640666. doi: 10.3389/fnins.2021.640666. eCollection 2021. PMID 33967678
- [Background] Woo SY, Joh JH, Han SA, Park HC. Prevalence and risk factors for atherosclerotic carotid stenosis and plaque: A population-based screening study. Medicine (Baltimore). 2017 Jan;96(4):e5999. doi: 10.1097/MD.0000000000005999. PMID 28121957
- [Background] Hackam DG. Optimal Medical Management of Asymptomatic Carotid Stenosis. Stroke. 2021 Jun;52(6):2191-2198. doi: 10.1161/STROKEAHA.120.033994. Epub 2021 May 5. PMID 33947208
- [Background] Kwapong WR, Liu J, Wan J, Tao W, Ye C, Wu B. Retinal Thickness Correlates with Cerebral Hemodynamic Changes in Patients with Carotid Artery Stenosis. Brain Sci. 2022 Jul 25;12(8):979. doi: 10.3390/brainsci12080979. PMID 35892420
- [Background] Song P, Fang Z, Wang H, Cai Y, Rahimi K, Zhu Y, Fowkes FGR, Fowkes FJI, Rudan I. Global and regional prevalence, burden, and risk factors for carotid atherosclerosis: a systematic review, meta-analysis, and modelling study. Lancet Glob Health. 2020 May;8(5):e721-e729. doi: 10.1016/S2214-109X(20)30117-0. PMID 32353319
- [Background] Cohen R, Padilla J, Light D, Diller R. Carotid artery occlusive disease and ocular manifestations: Importance of identifying patients at risk. Optometry. 2010 Jul;81(7):359-63. doi: 10.1016/j.optm.2009.10.013. PMID 20630374
- [Background] Batu Oto B, Kilicarslan O, Kayadibi Y, Yilmaz Cebi A, Adaletli I, Yildirim SR. Retinal Microvascular Changes in Internal Carotid Artery Stenosis. J Clin Med. 2023 Sep 16;12(18):6014. doi: 10.3390/jcm12186014. PMID 37762953
- [Background] Arthur A, Alexander A, Bal S, Sivadasan A, Aaron S. Ophthalmic masquerades of the atherosclerotic carotids. Indian J Ophthalmol. 2014 Apr;62(4):472-6. doi: 10.4103/0301-4738.121183. PMID 24817748
- [Background] Mursch-Edlmayr AS, Luft N, Podkowinski D, Ring M, Schmetterer L, Bolz M. Laser speckle flowgraphy derived characteristics of optic nerve head perfusion in normal tension glaucoma and healthy individuals: a Pilot study. Sci Rep. 2018 Mar 28;8(1):5343. doi: 10.1038/s41598-018-23149-0. PMID 29593269
- [Background] Luft N, Wozniak PA, Aschinger GC, Fondi K, Bata AM, Werkmeister RM, Schmidl D, Witkowska KJ, Bolz M, Garhofer G, Schmetterer L. Ocular Blood Flow Measurements in Healthy White Subjects Using Laser Speckle Flowgraphy. PLoS One. 2016 Dec 13;11(12):e0168190. doi: 10.1371/journal.pone.0168190. eCollection 2016. PMID 27959905
- [Background] Bissacco D, Attisani L, Settembrini AM, Fossati A, Carmo M, Dallatana R, Settembrini PG. Modifications in Near Infrared Spectroscopy for Cerebral Monitoring During Carotid Endarterectomy in Asymptomatic and Symptomatic Patients. Ann Vasc Surg. 2022 Feb;79:239-246. doi: 10.1016/j.avsg.2021.06.047. Epub 2021 Oct 10. PMID 34644636
- [Background] Ismail A, Chen HC, Faye I, Tang TB. Longitudinal effects of common carotid artery stenosis on ocular hemodynamics assessed using laser speckle flowgraphy in a rabbit model. Sci Rep. 2020 Sep 28;10(1):15829. doi: 10.1038/s41598-020-72556-9. PMID 32985560